CLINICAL TRIAL: NCT02875314
Title: HeadStart4: Newly Diagnosed Children (<10 y/o) With Medulloblastoma and Other CNS Embryonal Tumors Clinical and Molecular Risk-Tailored Intensive and Compressed Induction Chemotherapy Followed by Consolidation With Randomization to Either Single Cycle or to Three Tandem Cycles of Marrow-Ablative Chemotherapy With Autologous Hematopoietic Progenitor Cell Rescue
Brief Title: HeadStart4: Newly Diagnosed Children (<10 y/o) With Medulloblastoma and Other CNS Embryonal Tumors
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Parth Patel (Other)
Collaborators: Children's of Alabama (Other)
Responsible Party: Sponsor-Investigator, Parth Patel, Prinicipal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-00399
Record Dates: First submitted 2016-04-27; First posted 2016-08-23 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Medulloblastoma; Central Nervous System Embryonal Tumors
MeSH Terms: conditions — Medulloblastoma | interventions — Neoadjuvant Therapy; Vincristine; Cisplatin; Cyclophosphamide; Etoposide; Methotrexate; Carboplatin; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (3):
- Induction (Experimental): The 5 chemotherapy drugs used in the Induction part of treatment are vincristine, cisplatin, cyclophosphamide, etoposide and high-dose methotrexate.
  Three medications are also given to help reduce the side effects of the chemotherapy drugs. Filgrastim will be given through a vein or through a tiny needle into the tissue just under the skin to help blood counts recover after the chemotherapy. Mesna will be given through a vein with cyclophosphamide to help prevent bleeding in the bladder. Leucovorin will be given through a vein after the methotrexate to protect the body from the side effects of the methotrexate.
  Interventions: Drug: Induction
- Single Cycle Intensive Chemotherapy (Experimental): The three drugs to be used in this research study are thiotepa, etoposide and carboplatin. These drugs will be given over 6 days to help kill the cancer cells. After 72 hours from getting these drugs, previously collected and frozen blood cells will be thawed and returned through the venous catheter.
  Carboplatin is given by vein over 4 hours. Thiotepa is given by vein over 3 hours. Etoposide is given by vein over 3 hours. The schedule for these drugs is as follows:
  Day -8: Carboplatin Day -7: Carboplatin Day -6: Carboplatin Day -5: Thiotepa, Etoposide Day -4: Thiotepa, Etoposide Day -3: Thiotepa, Etoposide Day -2: Rest Day -1: Rest Day 0: Re-infusion of blood cells
  Interventions: Drug: Single Cycle Intensive Chemotherapy
- Tandem 3 Cycle Intensive Chemotherapy (Experimental): The 2 drugs to be used in this treatment are thiotepa and carboplatin. These drugs will be given over 2 days to help kill the cancer cells. After 72 hours from getting these drugs, previously collected and frozen blood cells will be thawed and returned through the venous catheter.
  Day -4: Thiotepa, Carboplatin Day -3: Thiotepa, Carboplatin Day -2: Rest Day -1: Rest Day 0: Re-infusion of blood cells.
  Following recovery from the first cycle of this chemotherapy, about 28 days following the Day 0 reinfusion of blood cells, the same cycle will be repeated again. A total of 3 cycles of this therapy will be administered, over the course of 12 weeks.
  Interventions: Drug: Tandem 3 Cycle Intensive Chemotherapy

INTERVENTIONS:
Drug: Induction — vincristine, cisplatin, cyclophosphamide, etoposide, high-dose methotrexate
  Other Names: vincristine, cisplatin, cyclophosphamide, etoposide, high-dose methotrexate
  Arms: Induction
Drug: Single Cycle Intensive Chemotherapy — Carboplatin, thiotepa, etoposide
  Other Names: Carboplatin, thiotepa, etoposide
  Arms: Single Cycle Intensive Chemotherapy
Drug: Tandem 3 Cycle Intensive Chemotherapy — Carboplatin, thiotepa
  Other Names: Carboplatin, thiotepa
  Arms: Tandem 3 Cycle Intensive Chemotherapy

SUMMARY:
This is a prospective randomized clinical trial, to determine whether dose-intensive tandem Consolidation, in a randomized comparison with single cycle Consolidation, provides an event-free survival (EFS) and overall survival (OS). The study population will be high-risk patients (non-Wnt and non-Shh sub-groups) with medulloblastoma, and for all patients with central nervous system (CNS) embryonal tumors completing "Head Start 4" Induction. This study will further determine whether the additional labor intensity (duration of hospitalizations and short-term and long-term morbidities) associated with the tandem treatment is justified by the improvement in outcome. It is expected that the tandem (3 cycles) Consolidation regimen will produce a superior outcome compared to the single cycle Consolidation, given the substantially higher dose intensity of the tandem regimen, without significant addition of either short-term or long-term morbidities.

DETAILED DESCRIPTION:
Due to the inferior response and event-free survival data of Regimens D and D2 on "Head Start III" for all children with supratentorial embryonal tumors, in comparison with the published data from "Head Start II" with Regimen A2 for metastatic patients, all such patients will receive the "Head Start II" Induction Regimen A2, on "Head Start 4", for either three or five cycles, depending upon whether or not they achieve complete remission by the end of Induction cycle #3. They will then undergo randomization to either single cycle or three tandem cycles of Consolidation marrow-ablative chemotherapy with AuHPCR.

Because of the unsatisfactory event-free survival for young children with non-desmoplastic/extensive nodular medulloblastoma (predominantly non-Shh and non-Wnt medulloblastoma subgroups) on Regimens D and D2 of "Head Start III", all these patients will receive the "Head Start II" Induction Regimen A2 on ""Head Start 4"", for either three or five cycles, depending upon whether or not they achieve complete remission by the end of Induction cycle #3. They will then undergo randomization to either single cycle or three tandem cycles of Consolidation marrow-ablative chemotherapy with AuHPCR.

Because of the excellent event-free and overall survival for young children with good risk medullo-blastoma (Shh or Wnt subgroups) treated with up-front "Head Start" chemotherapy strategies, such patients will undergo risk-tailored reduction of duration of Induction therapy from five cycles to three cycles of the "Head Start II" Induction Regimen A2 on "Head Start 4" for patients achieving a complete response to 3 cycles, followed, provided they are also without evidence of residual tumor following recovery from Induction cycle #3. They will NOT then undergo randomization, but will follow with a single cycle of Consolidation marrow-ablative chemotherapy as in "Head Start" studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 10 years of age at the time of definitive confirmatory eligible histologic or cytologic diagnosis of eligible CNS tumor (brain or spinal cord)
* Patients may not have received irradiation or chemotherapy (except corticosteroids)
* Have histologically proven diagnosis of medulloblastoma or CNS embryonal tumors of the brain or spinal cord
* Medulloblastoma

  * Posterior fossa classic, desmoplastic or extensive nodular or anaplastic/large cell medulloblastoma with appropriate and sufficient tumor material (FFPE or snap frozen) for proposed assays: all stages, age less than 6 years at diagnosis
  * Posterior fossa classic or anaplastic/large cell medulloblastoma with sufficient tumor material (FFPE or snap frozen) for proposed assays: clinically high-stage (neuraxis or extra-neural dissemination, M1-4), age greater than 6 years to less than 10 years at diagnosis
  * Posterior fossa medulloblastoma, those 6 years of age and above at diagnosis, will only be eligible if they have evidence of neuraxis or extraneural dissemination. Patients 6 years of age and above with low-stage (standard-risk, M0) medulloblastoma will NOT be eligible for this study, irrespective of molecular subgroup and extend of local resection
* CNS Embryonal Tumors:

  - Pineoblastoma, CNS neuroblastoma, CNS ganglioneuroblastoma, embryonal tumor with multi-layered rosettes (ETMR, including embryonal tumor with abundant neuropil and true rosettes (ETANTR), ependymoblastoma and ETMR not otherwise specified), medulloepithelioma, CNS embryonal tumor with rhabdoid features (INI1 intact) and CNS embryonal tumor, not otherwise specified.
* Must commence Induction chemotherapy within 28 days of the most recent definitive surgical procedure and within 21 days of the most recent neuro-imaging studies (MRI of brain, performed with and without gadolinium contrast, and MRI of total spine, performed with gadolinium contrast) and lumbar CSF cytological examination
* Patients must have adequate organ functions at the time of registration:

  * Liver: bilirubin less than 1.5 mg/dL (except for patients with Gilbert's Syndrome of indirect hyperbilirubinemia) and transaminases [SGPT or ALT, and SGOT or AST] less than 2.5 (two and a half) times the upper limits of institutional normal.
  * Renal: Creatinine clearance and/or glomerular filtration rate (GFR) greater than or equal to 60 mL/min/1.73m² within 21 days of protocol therapy.
  * Bone Marrow Function:

    1. Peripheral absolute phagocyte count (APC) > 1000/ µL. APC = numbers of banded neutrophils + segmented neutrophils + metamyelocytes + monocytes + eosinophils Please note, if institution reports differential as a percentage, then APC = [percentage of banded neutrophils + segmented neutrophils+ metamyelocytes+monocytes+eosinophils] x total white cell count.
    2. Platelet Count > 100,000/µL (transfusion independent)
    3. Hemoglobin > 8 gm/dL (may have received RBC transfusions).

Exclusion Criteria:

* Patients older than 10 years of age at time of diagnosis
* Following diagnoses are not eligible for study enrollment: CNS atypical teratoid/rhabdoid tumor (AT/RT); all ependymomas including anaplastic ependymomas of the brain or spinal cord; all choroid plexus carcinomas; all high-grade glial and glio-neuronal tumors; all primary CNS germ cell tumors; all primary CNS sarcomas; all primary or metastatic CNS lymphomas and solid leukemic lesions (i.e., chloromas, granulocytic sarcomas).
* Patients with unbiopsied diffuse intrinsic pontine tumors will NOT be eligible for this study.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Compare tandem consolidation vs. single cycle consolidation A | 5 years
  Dose-intensive tandem Consolidation will be compared with single cycle consolidation via randomization. The randomized consolidations will provide an event-free survival (EFS) analysis after completing "Head Start 4" Induction.
Compare tandem consolidation vs. single cycle consolidation B | 5 years
  Dose-intensive tandem Consolidation will be compared with single cycle consolidation via randomization. The randomized consolidations will provide an overall survival (OS) analysis after completing "Head Start 4" Induction.

SECONDARY OUTCOMES:
Induction Cycle Reduction | 5 years
  Induction chemotherapy cycles will be reduced in number from five to three for molecularly high-risk medulloblastoma (non-Shh/non-Wnt) and CNS embryonal tumors who achieve a complete response (CR) after three cycles of Induction therapy results in equivalent 3-year EFS. Outcome will be analyzed irrespective of Consolidation assignment (Primary Aim) and compared to historical controls.
Uniform Treatment Regimen | 5 years
  Assess the rate of response of sequential dose-intensive and dose-compressed Induction chemotherapy followed by marrow-ablative chemotherapy and autologous hematopoietic progenitor cell rescue (AuHPCR) for children with medulloblastoma and other CNS embryonal tumors enrolled on the "Head Start 4" study utilizing a uniform treatment regimen.
Therapy-Related Hearing Loss Evaluation A | 5 years
  The prevalence and severity of therapy-related hearing loss as a function of cumulative dosing of cisplatin (three versus five cycles during Induction) will be evaluated. Distortion-Product Oto-acoustic Emissions (DPOAE) will be used as an early predictor of hearing loss to identify at-risk patients.
Therapy-Related Hearing Loss Evaluation B | 5 years
  The prevalence and severity of therapy-related hearing loss as a function of AuHPCR (one versus three tandem transplants in Consolidation) will be evaluated. Distortion-Product Oto-acoustic Emissions (DPOAE) will be used as an early predictor of hearing loss to identify at-risk patients.
Neuropsychological effects will be evaluated using age based tests and questionnaires. | 5 years
  The long-term neuropsychological effects will be evaluated.
Endocrine studies will be conducted using Serum-free T4, TSH, Cortisol, IGF and IGFBP3 laboratory tests. | 5 years
  The long-term endocrine functions effect will be evaluated.
Physical growth will be evaluated by collecting patient's height, weight and BSA. | 5 years
  The long-term physical growth effect will be evaluated.
The development of second neoplasms will be monitored. | 5 years
  The long-term development of second neoplasms will be evaluated.
Neuropathology Biorepository and Clinical Database | 5 years
  The study will establish a "Head Start 4" repository of clinical, radiographic and biologic specimens, including nucleic acids derived from these specimens, for future genomic, biologic and pharmacologic research.

CONTACTS AND LOCATIONS:
Overall Officials: Randal Olshefski, MD, Principal Investigator — Nationwide Children's Hospital; Jonathan Finlay, MD, Study Chair — Global Neuro-Oncology, Inc.; Girish Dhall, MD, Study Chair — Children's of Alabama at UAB
Locations (62):
- United States (55):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Memorial Care Health Services, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital (UCLA), Los Angeles, California
  - UCSF Oakland Benioff, Oakland, California
  - Children's Hospital Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Center for Cancer and Blood Disorders, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Children's Hospital/ University of FL, Gainesville, Florida
  - Nemours Center for Cancer and Blood Disorders, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Orlando Health, Orlando, Florida
  - John's Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Children's Hospital/University of Indiana, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Louisville School of Medicine, Louisville, Kentucky
  - John's Hopkins University School of Medicine, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Central Michigan University, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital of Minnesota, Minneapolis, Minnesota
  - Masonic Children's Hospital/University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Specialty Care of Nevada, Las Vegas, Nevada
  - Joseph Sanzari Children's Hospital/ Hackensack University, Hackensack, New Jersey
  - Morristown Medical Center, Atlantic Health System, Morristown, New Jersey
  - New York Medical College, Hawthorne, New York
  - Northwell Health, Hempstead, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia Presbyterian Children's Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Golisano Children's Hospital/ SUNY Upstate Medical University, Syracuse, New York
  - Carolina's HealthCare System/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - American Family Children's Hospital/University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - B.C. Children's Hospital, Vancouver, British Columbia
  - Alberta Children's Hospital, Calgary
  - Stollery Children's Hospital, Edmonton
  - Hamilton Health/McMasters Children's Hospital, Hamilton, Canada, Hamilton
  - The Hospital of Sick Children, Toronto
- New Zealand (2):
  - Starship Children's Hospital, Auckland
  - Christchurch Children's Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: Undecided